CLINICAL TRIAL: NCT05043857
Title: Stereotactic PAncreatic RadioTherapy Adjuvant Therapy (SPARTA): Phase II Trial.
Brief Title: Stereotactic PAncreatic RadioTherapy Adjuvant Therapy
Acronym: SPARTA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2957
Record Dates: First submitted 2021-09-08; First posted 2021-09-14 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adjuvant Stereotactic Pancreatic Radiotherapy (Experimental): Postoperative Stereotactic Body Radiation Therapy (SBRT) after pancreatic tumor resection.
  Stereotactic Body Radiotherapy (SBRT) is a novel radiotherapy technique consisting of highly focused irradiation with a steep dose gradient, thus allowing the delivery of ablative radiation doses and significant sparing of proximity critical structures. Higher doses per fraction allows for more intensive treatments and shorter duration of the radiation course.
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy (SBRT) — Postoperative Stereotactic Body Radiation Therapy (SBRT) after tumor resection targeting 2 volumes
  * CTV1 (clips+isotropic 5mm expansion, edited on anatomic barriers): receiving 40 Gy in 5 fractions of 8 Gy
  * CTV2 (CTV1+ anisotropic 10-15 mm expansion including corresponding vessels, retroperitoneum posterior to the SMV/SMA or celiac axis, edited on anatomic barriers): receiving 30 Gy in 5 fractions of 6 Gy.

SUMMARY:
While surgery is considered the only potentially curative therapy for pancreatic cancer, 5-year overall survival (OS) is typically <25%. Following surgical resection of pancreatic cancer, adjuvant conventionally fractionated RT (CRT, delivering 45-54 Gy in 1.8-2.0 Gy per fraction) with 5-FU chemotherapy is recommended in high-risk patients (positive lymph nodes and/or R1-R2 resection margin status). However, the benefit of CRT in this setting is controversial due to lack of prospective positive data. Moreover, duration of treatment course (delaying initiation of more effective chemotherapy schedules), insufficient dose delivery due potential radiation-related severe toxicity to proximity organs represents a serious limitation to treatment efficacy. Stereotactic Body Radiotherapy (SBRT) is a novel radiotherapy technique consisting of highly focused irradiation with a steep dose gradient, thus allowing the delivery of ablative radiation doses and significant sparing of proximity critical structures. Higher doses per fraction allows for more intensive treatments and shorter duration of the radiation course.

DETAILED DESCRIPTION:
Pancreatic carcinoma is expected to become in the next 10 years the second leading cause of cancer-related mortality. Resection is the only treatment with the potential to achieve long-term survival, although expected survival at 5 year is <25%: postoperative use of local and systemic adjuvant treatments has been proposed to improve outcome While the efficacy of adjuvant chemotherapy, in parrticular multiagent chemotherapy, has been established, the potential impact of chemoradiation in the adjuvant setting is still controversial. However, its use in patients with high risk features such as nodal involvement and close or positive margins may be of interest.

Adjuvant chemoradiation, when clinically indicated, is usually delivered in a 6 week treatment course in association with concurrent dose-adapted chemotherapy, implying the necessity to interrupt more effective multi-agent chemotherapy schedules due to risk of increased toxicity.

It has been proposed that higher radiotherapy doses may result in improved outcome although a potential detrimental effect on survival of dose escalation >55 Gy with conventional fractionation, possibly related to increased toxicity, has been reported. Stereotactic Body Radiotherapy (SBRT) is a novel radiotherapy technique consisting of highly focused irradiation with a steep dose gradient, thus allowing the delivery of ablative radiation doses and significant sparing of proximity critical structures. Higher doses per fraction allows for more intensive treatments and shorter duration of the radiation course. In a retrospective study by Rwigema et al, adjuvant pancreatic SBRT was shown to be a safe and feasible treatment option for patients with high-risk pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Surgically treated T1-T4 adenocarcinoma with or without prior chemotherapy AND close (<2.5mm)/positive resection margin AND/OR N1 staging at lymphadenectomy
* ECOG performance status <2
* Age > 18
* Estimated life expectancy > 6 months
* Ability to provide written informed consent
* Cardiovascular comorbidities limiting life expectancy

Exclusion Criteria:

* Metastatic disease
* Biliary tract or neuroendocrine neuroplasm
* History of malignancies except for non-melanoma cutaneous tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Local Recurrence Rate | 1 year
  local recurrence rate in operated pancreatic cancer patients following adjuvant SBRT

SECONDARY OUTCOMES:
disease-free interval | 1 year
  disease-free interval in operated pancreatic cancer patients following adjuvant SBRT
Overall Survival | 1 year
  Overall Survival in operated pancreatic cancer patients following adjuvant SBRT

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Rozzano, MI, Italy

IPD SHARING:
Plan to Share IPD: No